CLINICAL TRIAL: NCT05893979
Title: Myopia Control Spectacle Lens Use Cessation Study
Brief Title: Myopia Control Spectacle Lens Cessation Study
Acronym: BIRCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPRO-2303-001
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-12

CONDITIONS: Myopia; Myopia Progression; Juvenile Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test Lens Group (Active Comparator)
  Interventions: Device: Spectacle Lenses
- Control Lens Group (Active Comparator)
  Interventions: Device: Spectacle Lenses

INTERVENTIONS:
Device: Spectacle Lenses — Standard Spectacle Lenses

SUMMARY:
To quantify myopic progression (cycloplegic spherical equivalent refraction - cSER) following the cessation of use of specific spectacle lenses.

To quantify axial length progression following cessation of use of specific spectacle lenses.

ELIGIBILITY:
Inclusion Criteria:

* Previously a successfully completed participant in the CYPRESS Extension study;
* Agree to wear the assigned spectacles constantly except for sleeping, swimming, or other activities in which spectacle wear would be dangerous or otherwise not possible (minimum of 10 hours per day);
* Willingness to participate in the trial for up to 12 months without contact lens wear;
* The subject's parent(s) or legal guardian(s) must read, understand, and sign the Statement of Informed Consent and receive a fully executed copy of the form.

Exclusion Criteria:

* Known allergy to proparacaine, tetracaine, or tropicamide.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic Spherical Equivalent Refraction (cSER) | 12 months
  Change in cSER

SECONDARY OUTCOMES:
Cycloplegic Spherical Equivalent Refraction (cSER) | 6 months
  Change in cSER
Axial Length (AL) | 12 months
  Change in AL

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Golden Optometric Group, Whittier, California
  - Omega Vision Center PA, Longwood, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Advanced Eyecare PC, Raytown, Missouri
  - Sacco Eye Group, Vestal, New York
  - Total Eye Care, Memphis, Tennessee
  - Vision Optique, Houston, Texas
  - William J Bogus, OD, FAAO, Salt Lake City, Utah